CLINICAL TRIAL: NCT00548184
Title: A Phase II Trial of Lapatinib and Trastuzumab With or Without Endocrine Therapy in Locally Advanced HER2 Overexpressing Breast Cancer Patients
Brief Title: Lapatinib and Trastuzumab With or Without Endocrine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-20464
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: primary breast cancers; Locally advanced breast cancers
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group Assignment (Experimental): Lapatinib Trastuzumab Endocrine
  Interventions: Drug: Lapatinib; Drug: Trastuzumab; Drug: Endocrine

INTERVENTIONS:
Drug: Lapatinib — Monoclonal Antibody
  Other Names: TyKerb
Drug: Trastuzumab — Monoclonal Antibody
  Other Names: Herceptin
Drug: Endocrine — Hormonal Therapy
  Other Names: Varies

SUMMARY:
We think that lapatinib will help to shrink your tumor when given prior to the main or primary therapy for the kind of breast cancer you have been diagnosed with. When treatment is given before the main or primary therapy, it is called neoadjuvant therapy. We will compare lapatinib with lapatinib plus trastuzumab (herceptin) for 12 weeks. If your tumor is estrogen receptor positive (ER positive), estrogen deprivation will also be given to you. Tumors that are ER positive have a lot of estrogen receptors found in them. This is also called "over expression" or amplification of estrogen receptors.

The most important information we will get from this study is to see the response to "neoadjuvant" (treatment given before the main treatment), lapatinib with trastuzumab (herceptin) in your tumor tissue sample.

DETAILED DESCRIPTION:
The neoadjuvant setting is especially attractive for studies of predictive biologic correlates for several reasons including early assessment of response to therapy, access to the primary tumor, and reduced patient numbers compared to those required in the adjuvant setting. Response to neoadjuvant therapy is a validated surrogate marker for improved survival; it may be used to test the overall efficacy of neoadjuvant treatment regimens and response in the primary tumor mirrors the effect of therapy on micrometastases.

Trastuzumab is an efficacious agent in HER2 overexpressing breast cancers. Our results with neoadjuvant trastuzumab indicate that its efficacy may be better in patients with treatment-naïve tumors compared to metastatic disease, with 26% of patients showing a partial response after only 3 weeks of therapy. No patients progressed during this 3-week period. We have also conducted a neoadjuvant lapatinib study given as a single agent for 6 weeks. The response rates in this second study have been impressive with greater than 80% responses in patients with HER2 positive locally advanced breast cancers. It is likely that the true response rate to HER2 blockade would be higher had therapy been continued for longer. We therefore hypothesize that lapatinib, a dual tyrosine kinase inhibitor, together with trastuzumab, will result in tumor regression when given as neoadjuvant therapy in HER2 overexpressing breast cancer. We will compare lapatinib plus trastuzumab for 12 weeks, and if the tumors express ER, estrogen deprivation will also be administered.

This is a phase II trial. Clinical efficacy will be assessed by bidimensional tumor measurements of the primary cancer at baseline, and at the end of week 12. Objective tumor response rate defined as objective bidimensional tumor measurements after neoadjuvant treatment at 12 weeks will be calculated, and assessed according to standard RECIST criteria. Pathologic responses will be graded as pathologic complete response if there is no invasive cancer in the residual breast at the time of surgery. Near pathologic complete response will also be documented as residual disease of less than 1 cm.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be female.
* Signed informed consent.
* Locally advanced breast cancers or primary breast cancers are eligible. Locally advanced cancers must be of clinical and/or radiologic size >3 cm, or >2 cm with clinical evidence of axillary nodal involvement. (If tumors are less than 3 cm, we will use radiologically measured tumor size to determine the minimal tumor size for eligibility and in assessing tumor size during follow-up).
* HER2 overexpressing tumors defined as HercepTest score of 3+, or > 10% cells moderately or strongly HER2 positive by other methods, or Allred semi-quantitative score of >5, or gene amplified.
* Negative serum pregnancy test (HCG) within 7 days of starting study, if of child-bearing potential.
* Kidney and liver function tests - all within 1.5 times the institution's upper limit of normal.
* Performance status (WHO scale) less than 2 and life expectancy more than 6 months.
* Age at least 18 years.
* No brain or leptomeningeal disease.
* No previous or current malignancies at other sites within the last 5 years, with exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.

Note: The presence of pathological involvement of axillary nodes will be assessed and agreed upon by two investigators.

Exclusion Criteria:

* Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
* Severe underlying chronic illness or disease.
* Cardiomyopathy or baseline LVEF less than 50%.
* Other investigational drugs while on study.
* Severe or uncontrolled hypertension, history of congestive heart failure or severe coronary arterial disease.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded
* Taking any lapatinib-prohibited medication within 7 days of first dose of study medications. (See Prohibited Medications List in protocol.)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (6):
- United States (6):
  - UAB Cancer Center, Birmingham, Alabama
  - The University of Chicago, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Bunting-Blaustein Cancer Research, Baltimore, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Lester and Sue Smith Breast Center, Houston, Texas

REFERENCES:
- [Derived] Veeraraghavan J, De Angelis C, Mao R, Wang T, Herrera S, Pavlick AC, Contreras A, Nuciforo P, Mayer IA, Forero A, Nanda R, Goetz MP, Chang JC, Wolff AC, Krop IE, Fuqua SAW, Prat A, Hilsenbeck SG, Weigelt B, Reis-Filho JS, Gutierrez C, Osborne CK, Rimawi MF, Schiff R. A combinatorial biomarker predicts pathologic complete response to neoadjuvant lapatinib and trastuzumab without chemotherapy in patients with HER2+ breast cancer. Ann Oncol. 2019 Jun 1;30(6):927-933. doi: 10.1093/annonc/mdz076. PMID 30903140
- [Derived] Rimawi MF, Mayer IA, Forero A, Nanda R, Goetz MP, Rodriguez AA, Pavlick AC, Wang T, Hilsenbeck SG, Gutierrez C, Schiff R, Osborne CK, Chang JC. Multicenter phase II study of neoadjuvant lapatinib and trastuzumab with hormonal therapy and without chemotherapy in patients with human epidermal growth factor receptor 2-overexpressing breast cancer: TBCRC 006. J Clin Oncol. 2013 May 10;31(14):1726-31. doi: 10.1200/JCO.2012.44.8027. Epub 2013 Apr 8. PMID 23569315

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib + Trastuzumab: All study participants received lapatinib 1000mg daily and Trastuzumab 4mg/kg loading dose and then 2mg/kg every week
Period: Overall Study
Arm/Group | Lapatinib + Trastuzumab
Started | 65
Completed | 60 (65 patients were on treatment. 5 did not complete due to adverse events or other reasons.)
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — took other drug | 1
Not completed — Found Her2 negative | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib + Trastuzumab
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 49 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Assessment After Study Treatment
Description: Pathologic Assessment After 12 weeks of lapatinib and trastuzumab with or without endocrine therapy. Pathologic complete response: no invasive cancer in the residual breast. Near pathologic complete response: residual disease of less than 1 cm in breast.
Time Frame: 12 weeks
Population: 65 patients were enrolled and received the study treatment. 1 patient was found ineligible for this study therefore she was excluded from outcome report.
Measure: Number; unit: participants
Groups:
- Lapatinib + Trastuzumab: All study participants received lapatinib 1000mg daily and trauzumab 4mg/kg loading dose and then 2mg/kg every week
Arm/Group | Lapatinib + Trastuzumab
Number analyzed (Participants) | 64
participants
  Complete Pathologic Response | 18
  Near Complete Pathologic Response | 16
  Not Pathologic response | 30

2. Other Pre Specified Outcome: Data Analysis of the Biomarkers: Immunohistochemical Staining of Cells From Breast Biopsies and Skin Biopsies Will be Performed.
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: study treatment up to 12 weeks
Arm/Group | Lapatinib + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 2/65
Other Adverse Events (participants affected / at risk) | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Trastuzumab (N=65)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib + Trastuzumab (N=65)
ALT, SGPT (Metabolism and nutrition disorders) | 15 (19)
AST, SGOT (Metabolism and nutrition disorders) | 12 (18)
Alkaline phosphatase (Metabolism and nutrition disorders) | 7 (10)
Allergic reaction/hypersensitivity (Immune system disorders) | 4 (4)
Allergic rhinitis (Immune system disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 4 (4)
Bilirubin (Metabolism and nutrition disorders) | 5 (9)
Calcium, serum-low (Metabolism and nutrition disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 43 (55)
Dry Skin (Skin and subcutaneous tissue disorders) | 12 (12)
Fatigue (General disorders) | 21 (21)
Glucose, serum-high (Metabolism and nutrition disorders) | 11 (18)
HEARTBURN (Gastrointestinal disorders) | 12 (12)
HEMOGLOBIN (Blood and lymphatic system disorders) | 14 (19)
Hot flashes/flushes (Endocrine disorders) | 10 (10)
Hypertension (Cardiac disorders) | 7 (7)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 6 (6)
Insomnia (General disorders) | 7 (7)
Mood alteration (Nervous system disorders) | 8 (8)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 8 (8)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 20 (20)
pain (General disorders) | 10 (13)
Potassium, serum-low (Metabolism and nutrition disorders) | 13 (18)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 9 (13)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 30 (35)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (8)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes